CLINICAL TRIAL: NCT06559527
Title: Investigation of Pharmacokinetics, Safety and Tolerability of a Single Subcutaneous Dose of NNC0487-0111 in Participants With Various Degrees of Renal Impairment and Normal Renal Function
Brief Title: A Research Study Looking Into Blood Levels of the Medicine NNC0487-0111 in the Body and How Well it is Tolerated in Participants With Reduced Kidney Function and Normal Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9490-7611; U1111-1298-6886 (Other: World Health Organization (WHO)); 2023-509961-19 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Mild Renal Impairment (Experimental): Participants with mild renal impairment (estimated glomerular filtration rate [eGFR] - 60 - 89 milliliter per min [mL/min]) will administer a single dose of NNC0487-0111 on Day 1.
  Interventions: Drug: NNC0487-0111
- Moderate Renal Impairment (Experimental): Participants with moderate renal impairment (eGFR - 30 - 59 mL/min) will administer a single dose of NNC0487-0111 on Day 1.
  Interventions: Drug: NNC0487-0111
- Severe Renal Impairment (Experimental): Participants with severe renal impairment (eGFR - less than 30 mL/min not requiring dialysis) will administer a single dose of NNC0487-0111 on Day 1.
  Interventions: Drug: NNC0487-0111
- End-Stage Renal Disease (ESRD) (Experimental): Participants with ESRD (requiring dialysis treatment) will administer a single dose of NNC0487-0111 on Day 1.
  Interventions: Drug: NNC0487-0111
- Normal Renal Function (Experimental): Participants with normal renal function (eGFR - greater than or equals 90) will administer a single dose of NNC0487-0111 on Day 1.
  Interventions: Drug: NNC0487-0111

INTERVENTIONS:
Drug: NNC0487-0111 — Participants will administer a single dose of NNC0487-0111 subcutaneously using NovoPen®4 by injection into a skinfold on the abdomen.

SUMMARY:
Novo Nordisk is developing the study medicine NNC0487-0111 to treat people living with type 2 diabetes and/or people living with overweight or obesity. The aim of this study is to see if blood levels of NNC0487-0111 are the same in people living with various degrees of reduced kidney function as for people with normal kidney function. Participants will be given one single injection by the study staff in a skinfold in their stomach using a pen device (NovoPen®4).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-80 years (both inclusive) at the time of signing the informed consent
* Body mass index (BMI) between 20.0 and 39.9 kilogram per square meter (kg/m^2) (both inclusive) at screening.
* Meeting the pre-defined eGFR values based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation (2021) adjusted for the estimated individual body surface area (BSA);

  * Normal renal function - greater than or equal to 90 mL/min
  * Mild renal impairment - 60 - 89 (mL/min)
  * Moderate renal impairment - 30 - 59 (mL/min)
  * Severe renal impairment - less than 30 (mL/min) not requiring dialysis
  * End-stage renal disease (ESRD) - Requiring dialysis treatment
* For ESRD: Participants requiring dialysis treatment should be on current treatment with haemodialysis.

Exclusion Criteria:

* Any disorder, unwillingness, or inability which in the investigator's opinion might jeopardize participant's safety or compliance with the protocol.
* Use of drugs known to affect creatinine clearance including cephalosporin and aminoglycoside, antibiotics, flucytosine, cisplatin, cimetidine, trimethoprim, cibenzoline, and nitrofurantoin within 14 days or 5 half-lives, whichever is greater, before dosing the investigational medicinal product (IMP).
* Presence or history of any clinically relevant respiratory, metabolic, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions(except conditions associated with renal impairment or ESRD).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
AUC0111,0-∞,SD: Area under the NNC0487-0111 plasma concentration-time curve from time 0 to infinity after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of study visit (Visit 9, Day 28)
  Measured as hours*nanomole per liter (h*nmol/L).

SECONDARY OUTCOMES:
Cmax,0111,SD: Maximum observed plasma NNC0487-0111concentration after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of study visit (Visit 9, Day 28)
  Measured as nanomole per liter (nmol/L).
tmax,0111,SD: Time to maximum observed plasma NNC0487-0111 concentration after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of study visit (Visit 9, Day 28)
  Measured as hours.
t½,0111,SD: Terminal half-life of NNC0487-0111 after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of study visit (Visit 9, Day 28)
  Measured as hours.
Vz/F0111,SD: Apparent volume of distribution of NNC0487-0111 after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of study visit (Visit 9, Day 28)
  Measured as liter (L)
CL/F0111,SD: Apparent clearance of NNC0487-0111 after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of study visit (Visit 9, Day 28)
  Measured as liter per hour (L/h).
Number of treatment emergent adverse events (TEAEs) | From time of trial product administration (Visit 2, Day 1) until completion of the end of study visit (Visit 9, Day 28)
  Measured as number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com